CLINICAL TRIAL: NCT00463931
Title: Using Community-Based Volunteers to Reach Non-Enrolled School-Aged Children Through Community-Directed Treatment of Schistosomiasis in School-Aged Children in Rural Northern Ghana
Brief Title: Using Community-Based Volunteers to Reach Non-Enrolled School Aged Children Through Community-Directed Treatment of Schistosomiasis in School-Aged Children in Rural Northern Ghana
Status: Completed | Type: Observational
Sponsor: DBL -Institute for Health Research and Development (Other)
Other Study IDs: SRP-GH-FA-06
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: Schistosomiasis; Soil-Transmitted Helminthiasis
Keywords: Schistosomiasis; Soiltransmitted helminthiasis; Community-based volunteer; School based treatment approach
MeSH Terms: conditions — Schistosomiasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Schistosomiasis and soil-transmitted helminhtiasis occur throughout the developing world and are most prevalent in the poorest communitites. These worms have been linked to several nutritional and intellectual deficiencies in many endemic populations worldwide. Helminth control, though crucial has been neglected for varied reasons. Currently, interests towards the control of neglected diseases including schistosomiasis and soil-transmitted helminths has been revived through many interventions including repeated chemotherapy to help improve public health outcomes and prevent long term morbidity. This will contribute to achieving several of the Millennium Development Goals at a favourable cost. A community-directed treatment of human schistosomiasis and STH in school-aged children in rural notrhern Ghana using praziquantel and albendazole is proposed. It is planned to test the hypothesis that community-based volunteers are non-inferior and more cost effective than rural school teachers at reaching school-aged children.

DETAILED DESCRIPTION:
The primary objectives of the study are:

To compare coverage rate of community based volunteers and rural school teachers in the distribution of praziquantel and albendazole to scholl-aged children To determine the cost effectiveness of using community based volunteers to distribute praziquantel and albendazole to school-aged children in rural Ghana.

Study methods:

A list of all school-aged children (6-15 years) in the study area will be generated from the Navrongo Demographic Surveillance System database and registers produced and given to all school teachers and community based volunteers who will be responsible for the distribution of the antihelminithics. The school teachers and community based volunteers will provide the drugs to both enrolled and non-enrolled school-aged children. Percentage coverage of school-aged children will be the outcome measure and compated between the school teachers and the community based volunteers. Stool and urine samples will be collected from a representative sample (916) of the children for laboratory analysis before the administration of the drugs for baseline data. Sample collection and laboratory analysis will be repeated 6 and 12 months after the first round of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Children between 6 and 15 years of age

Ages: 6 Years to 15 Years | Sex: All
Age Groups: Child
Enrollment: 916
Dates: Start 2006-09; Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis Anto, MD, Principal Investigator — Navrongo Health Research Centre, Ghana
Locations (1):
- The Navrongo Health Research Centre, Navrongo, Ghana